CLINICAL TRIAL: NCT05544617
Title: Recurrent Collection By Medical Student From Sorbonne-Université in General Medicine
Brief Title: Recurrent Collection By Medical Student in General Medicine
Acronym: RCIMG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sorbonne University (Other)
Responsible Party: Principal Investigator, Guillaume Avenin, Principal Investigator, Sorbonne University
Other Study IDs: 1
Record Dates: First submitted 2022-09-08; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: General Practice
Keywords: citizen science; Medical student; ICPC

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The project for the recurrent collection of data from interns in general medicine is a formalized description of the consultations attended by medical students during their outpatient training. This formalization uses the International Classification of Primary Care. This project aims to create a research network between general medical interns, mainly for their thesis, which pools their observations in a database accessible to all participants.

ELIGIBILITY:
Inclusion Criteria:

* consultation of his general practitioner

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: iterations of group of 5 consecutive patients consulting a general practice, regardless of the reason for consultation
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
reason for consultation | through study completion, an average of 6 month
  ICPC
diagnosis | through study completion, an average of 6 month
  ICPC

CONTACTS AND LOCATIONS:
Locations (1):
- guillaume AVENIN, Avon, France

IPD SHARING:
Plan to Share IPD: No